CLINICAL TRIAL: NCT07280104
Title: Investigation of Development Infants With Primary Congenital Hypothyroidism
Brief Title: Infants With Primary Congenital Hypothyroidism and Development
Status: Recruiting | Type: Observational
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Rabia ZORLULAR, principal investigator, Nigde Omer Halisdemir University
Other Study IDs: Congenital hypothyroidism
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Congenital Hypothyroidism
Keywords: Hypothyroidism; neurological status; motor development; sensory processing
MeSH Terms: conditions — Congenital Hypothyroidism; Hypothyroidism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- congenital hypothyroidism: The thyroid gland is responsible for producing hormones necessary for normal growth and development. Congenital hypothyroidism is a condition characterized by an underactive or absent thyroid gland in infants.
  Interventions: Behavioral: neurological status; Behavioral: sensory processing functions; Behavioral: Motor development
- Control Group: A control group of 20 healthy children, born at term and aged between 6 and 18 months, without primary congenital hypothyroidism will be created.
  Interventions: Behavioral: neurological status; Behavioral: sensory processing functions; Behavioral: Motor development

INTERVENTIONS:
Behavioral: neurological status — The Hammersmith Infant Neurological Examination (HINE) was planned to be used to assess the neurological status of infants. The HIND is a standardized examination for children aged 3 to 24 months, with high predictive value in the early detection of neurological disorders.
Behavioral: sensory processing functions — The Test of Sensory Function in Infants (TSFI) was planned to be used to assess infant sensory development. The TSFI is frequently used to assess the sensory processing functions of infants aged 4-18
Behavioral: Motor development — The Peabody Developmental Motor Scales-2 (PDMS-2) was planned to be used to assess motor development. The test is designed to identify developmental delays in children aged 0-72 months.

SUMMARY:
A review of the literature has focused primarily on the cognitive and motor development of children with congenital hypothyroidism, but no studies on sensory processing skills have been found. Considering the age range of the groups studied, studies conducted in the early stages of life are rare. This planned study aims to examine the neurological status, motor development, and sensory processing skills of infants aged 6-18 months, considering early synaptogenesis.

DETAILED DESCRIPTION:
The thyroid gland is responsible for producing the hormones necessary for normal growth and development. Congenital hypothyroidism is a condition characterized by underactive or absent thyroid gland in infants. Because thyroid hormone is essential for brain development, these children are at risk for brain damage and related cognitive and motor deficits. Initiating thyroxine supplementation early after birth through newborn screening programs aims to minimize this brain damage. Various studies on the effectiveness of these screening programs have shown that early thyroxine supplementation results in intelligence quotients within the normal range. However, mild cognitive and motor deficits, such as attention and balance problems, are present in most patients.

This planned study aims to examine the neurological status, motor development, and sensory processing skills in infants aged 6-18 months. The results of this study may provide a scientific basis for early follow-up and intervention programs by demonstrating the potential impact of congenital hypothyroidism on these developmental areas.

ELIGIBILITY:
Inclusion Criteria:

* Those with primary congenital hypothyroidism who have been treated since the newborn period and are currently on treatment.
* Infants born at term.
* Between 6 and 18 months old.

Exclusion Criteria:

* Infants with secondary congenital hypothyroidism,
* Preterm infants,
* Those with congenital infections or proven genetic alterations,
* Infants diagnosed with metabolic, neurological, or genetic diseases,
* Infants whose parents did not volunteer for the study

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Primary congenital hypothyroidism is an endocrine disorder that develops from birth due to insufficient thyroid hormone production by the thyroid gland. The term "primary" indicates that the problem originates directly from the thyroid gland itself, meaning there is no disorder at the hypothalamus or pituitary level. The study aims to recruit infants with and without primary congenital hypothyroidism (controls) who meet the inclusion criteria and whose parents provide voluntary consent.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-12-20 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Motor development | 6-18 month
  The Peabody Developmental Motor Scales-2 (PDMS-2) was planned to be used to assess motor development. The test is designed to identify developmental delays in children aged 0-72 months. Separate tests and rating scales are used to assess children's motor development, including both gross and fine motor skills. Each item in the PDMS-2 is scored on a 3-point ordinal scale reflecting the child's performance:
  2 points - the child performs the item according to the specified criteria;
  1 point - the child's performance shows emerging skill or partial success; 0 points - the child cannot or will not attempt the item, or the attempt does not meet criteria.
Sensory development | 6-18 months
  The Test of Sensory Functions in Infants (TSFI) was planned to be used to assess infant sensory development. The TSFI is frequently used to assess the sensory processing functions of infants aged 4-18 months. It is used to determine whether an infant has a sensory processing problem and to what extent. It consists of 24 items. The TSFI requires the infant to be stimulated and interact with various materials. The total score ranges from 0-49, and the test has normative values for different age groups. Although it is used from the fourth month onward, the most reliable and valid results are obtained between 7-18 months.
Neurological Examination | 6-18 months
  The Hammersmith Infant Neurological Examination (HINE) was planned to be used to assess the neurological status of infants. The HINE is a standardized examination for children aged 3 to 24 months, with high predictive value in the early detection of neurological disorders. It is a standardized clinical assessment tool developed to assess the neurological integrity, nervous system maturity, and potential neuromotor disorders in newborns. The HINE is grouped under three main subheadings: neurological, motor, and behavioral. Each item is scored from 0 to 3. The total score reflects the level of neurological maturity and abnormality. There are 26 items in total, with a maximum score of 78. A higher score indicates a more mature neurological status.

CONTACTS AND LOCATIONS:
Locations (1):
- Nigde Omer Halisdemir University, Niğde, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Naafs JC, Marchal JP, Fliers E, Verkerk PH, Luijten MAJ, Boelen A, van Trotsenburg ASP, Zwaveling-Soonawala N. Cognitive and Motor Outcome in Patients with Early-Detected Central Congenital Hypothyroidism Compared with Siblings. J Clin Endocrinol Metab. 2021 Mar 8;106(3):e1231-e1239. doi: 10.1210/clinem/dgaa901. PMID 33274354